CLINICAL TRIAL: NCT02971618
Title: Observational Retrospective Multicenter Study to Evaluate Clinical Outcome Variables Change With dapaGLiflozin Treatment Introduced in Patients With T2D uncOntrolled by the Current Therapy in Real Clinical Practice in RussIA
Brief Title: Study With Dapagliflozin
Acronym: GLORIA
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D1690R00030
Record Dates: First submitted 2016-11-21; First posted 2016-11-23 (Estimated); Last update posted 2019-08-06 (Actual); Status verified 2019-08

CONDITIONS: Diabetes Mellitus Type 2
Keywords: dapagliflozin,; Russia,; retrospective study,; diabetes mellitus type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Total group: Patients T2D with dapagliflozin treatment

SUMMARY:
The study will retrospectively collect clinical variables and socio-demographic data from medical records of patients with T2DM initiating treatment with dapagliflozin after the previous failure/inefficiency of other treatment options (defined as non-achievement of target Hb1Ac) and according to the officially approved indication as per instruction for the use of medicinal product.

It is expected that the best available data regarding clinical variables and patient socio-demographic profiled will be collected from the patient medical records at up to 40 major Russian outpatient clinics/centers specialized in the treatment and management of T2DM patients.

There are 2 time points:

* Baseline data: baseline data are defined as data available within 3 months prior to the first dose of dapagliflozin. In case of presence of multiple data values within baseline period the most recent pre-dose value will be selected
* Follow-up data: any post-baseline data will be considered as follow-up but the primary analysis will be focused on data available at 6 plus/minus 3 months after the initiation of dapagliflozin. In case of discontinuation dapagliflozin, data will be collected at routine visit within 3-month time frame after the last dose

DETAILED DESCRIPTION:
Objectives and Hypotheses:

Primary objective:

To describe HbA1c (glycosylated haemoglobin) change from baseline to follow-up

Secondary objectives:

Clinical data:

* To estimate percentage (%) of patients with reduction of HbA1c by 0.5% or more from baseline to follow-up
* To estimate percentage (%) of patients reaching the therapeutic glycemic response (HbA1c <7.0%) from baseline to follow-up
* To describe change of fasting blood glucose from baseline to follow-up
* To estimate change of body weight from baseline to follow-up
* To estimate percentage (%) of patients with body weight reduction by at least 5% from baseline to follow-up
* To estimate percentage (%) of patients with reduction of HbA1c by 0.5% or more and body weight reduction by at least 5% from baseline to follow-up
* To describe change of systolic and diastolic blood pressure from baseline to follow-up (systolic and diastolic, in mmHg)

Methods:

Study design:

The study will retrospectively collect clinical variables and socio-demographic data from medical records of patients with T2DM initiating treatment with dapagliflozin after the previous failure/inefficiency of other treatment options (defined as non-achievement of target Hb1Ac) and according to the officially approved indication as per instruction for the use of medicinal product.

It is expected that the best available data regarding clinical variables and patient socio-demographic profiled will be collected from the patient medical records at up to 40 major Russian outpatient clinics/centers specialized in the treatment and management of T2DM patients.

There are 2 time points:

* Baseline data: baseline data are defined as data available within 3 months prior to the first dose of dapagliflozin. In case of presence of multiple data values within baseline period the most recent pre-dose value will be selected
* Follow-up data: any post-baseline data will be considered as follow-up but the primary analysis will be focused on data available at 6 plus/minus 3 months after the initiation of dapagliflozin. In case of discontinuation dapagliflozin, data will be collected at routine visit within 3-month time frame after the last dose.

Data Source(s):

Participating investigators should be physicians-endocrinologists working in approximately 12 outpatient clinics specialized in management of patients with T2DM in Moscow. There is no current legislation on EMR in Russia, so, paper medical records will be utilized, and data collection using electronic CRFs will be done.

Study Population:

T2DM patients previously uncontrolled on standard therapy (mono-, double therapy with OADs: metformin, SU or DPP-4 inhibitors or on insulin) initiating treatment with dapagliflozin as monotherapy, combination with OADs or as add-on to insulin with available data on Hb1c within 3 months prior to the first dose of dapagliflozin. All consecutive patients at the clinic in inclusion period who meet inclusion and exclusion criteria will be included.

Exposure(s):

Only patients initiating treatment with dapagliflozin as monotherapy, combination with OADs or as add-on to insulin will be included in the study.

Outcome(s):

Population parameters

* Date of birth
* Gender
* Level of education
* Level of income
* Ethnicity/race
* Living conditions
* Working conditions All documented macro- and microvascular T2DM complications and concomitant medications (antidiabetic drugs, statins, ACE inhibitors, sartans, beta-blockers, calcium channel antagonists) will be collected for whole course of dapagliflozin administration.

Clinical parameters

* Hb1Ac
* Fasting glucose
* Body weight
* Blood pressure (systolic and diastolic)

Sample Size Estimations:

Approximate sample size is 850 patients.

Statistical Analysis:

Epidemiological methods mainly will be used to represent the study data. A descriptive analysis approach will be used to analyse study objectives. Descriptive statistics will be used to analyse the study population, baseline data and clinical outcomes. The descriptive statistics will include mean, standard deviation, median, minimum and maximum, range, number of valid cases for continuous variables, number, percentage, and distribution for categorical variables. The percentage will be given with the relevant two-sided 95% confidence intervals.

Only available data will be analyzed; no missing values imputation will be applied. Only patients with available data on HbA1c both within 3 months prior to the first dose of dapagliflozin and at 6±3 months after the initiation of dapagliflozin will be included in the main analysis.

All other baseline, effectiveness parameters will be tabulated, assessed in subgroups where available..

In order to evaluate the association between achievement of the HbA1C goals and patient characteristics, the multivariate logistic regression model was developed. A binary categorical attribute-HbA1C within/outside < 7% at 6±3 months after the initiation of dapagliflozin -serves as a dependable variable in this model

ELIGIBILITY:
Inclusion Criteria:

Patients with Type 2 Diabetes Mellitus Male and female, age 18-65 years (both inclusive) Patients with T2DM given a first prescription for dapagliflozin after Dec 2014 till 1 October 2016

Exclusion Criteria:

Type 1 diabetes Contraindications for SGLT 2 inhibitors (high individual sensitivity to SGLT 2 inhibitors, T1DM, diabetic ketoacidosis, moderate and severe renal failure (eGFR < 60 ml/min/1.73 m3), end-stage renal disease, lactose intolerance, intolerance of glucose and galactose, pregnancy and breast feeding, age younger than 18 years old, use of loop diuretics, decrease of circulating blood volume due to acute disease, age of 77 years old and older Prior use of SGLT 2 inhibitors

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: T2DM patients previously uncontrolled on standard therapy (mono-, double therapy with OADs: metformin, SU or DPP-4 inhibitors or on insulin) initiating treatment with dapagliflozin as monotherapy, combination with OADs or as add-on to insulin with available data on Hb1c within 3 months prior to the first dose of dapagliflozin. All consecutive patients at the clinic in inclusion period who meet inclusion and exclusion criteria will be included.
Sampling Method: Non-Probability Sample
Enrollment: 929 (Actual)
Dates: Start 2017-02-21 (Actual); Primary Completion 2018-08-03 (Actual); Study Completion 2018-08-03 (Actual)

PRIMARY OUTCOMES:
HbA1c (glycosylated haemoglobin) | 3 months
  To describe HbA1c (glycosylated haemoglobin) change from baseline to follow-up

SECONDARY OUTCOMES:
reduction of HbA1c by 0.5% or more | 3 months
  To estimate percentage (%) of patients with reduction of HbA1c by 0.5% or more from baseline to follow-up
(%) of patients reaching the therapeutic glycemic response (HbA1c <7.0%) | 3 months
  To estimate percentage (%) of patients reaching the therapeutic glycemic response (HbA1c <7.0%) from baseline to follow-up
change of fasting blood glucose | 3 months
  To describe change of fasting blood glucose from baseline to follow-up
change of body weight | 3 months
  To estimate change of body weight from baseline to follow-up
percentage (%) of patients with body weight reduction by at least 5% | 3 months
  To estimate percentage (%) of patients with body weight reduction by at least 5% from baseline to follow-up
percentage (%) of patients with reduction of HbA1c by 0.5% or more and body weight reduction by at least 5% | 3 months
  To estimate percentage (%) of patients with reduction of HbA1c by 0.5% or more and body weight reduction by at least 5% from baseline to follow-up
change of systolic and diastolic blood pressure | 3 months
  To describe change of systolic and diastolic blood pressure from baseline to follow-up (systolic and diastolic, in mmHg)

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir Bulatov, Study Director — AstraZeneca; Mikhail Antsiferov, Prof., Principal Investigator — Moscow endocrinology dispensary
Locations (2):
- Russia (2):
  - Research Site, Moscow
  - Research Site, Saint Petersburg

REFERENCES:
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D1690R00030&attachmentIdentifier=74eb5465-b987-433b-a09b-ee6ea1f2791c&fileName=GLORIA-CSR-SYNOPSIS_ENG.pdf&versionIdentifier=